CLINICAL TRIAL: NCT02268071
Title: Arrêt du Traitement Antihypertenseur Chez Les Patients Hypertendus Suivis en Médecine Générale / Stopping Antihypertensive Treatment amOng Hypertensive Patients in Primary Care: The STOP-Trial
Brief Title: Stopping Antihypertensive Treatment amOng Hypertensive Patients in Primary Care (STOP-Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Marc BOIVIN, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-001773-14
Record Dates: First submitted 2014-10-14; First posted 2014-10-20 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Hypertension
Keywords: Hypertension; Stopping antihypertensive treatment; Primary care; White coat hypertension; Masked Hypertension
MeSH Terms: conditions — Hypertension; White Coat Hypertension; Masked Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypertensive patients (Experimental): Antihypertensive treatment will be stopped for 1 year unless hypertension recurrence
  Interventions: Drug: Antihypertensive treatment will be stopped for 1 year unless hypertension recurrence

INTERVENTIONS:
Drug: Antihypertensive treatment will be stopped for 1 year unless hypertension recurrence — For patients with average of HBPM values <135/85mmHg at baseline, the antihypertensive treatment will be stopped for 1 year (half dose for 3 days then interruption)

SUMMARY:
The STOP-Trial is a prospective multicenter nonrandomized open study on grade I hypertension, performed by General practitioners.

The study will be conducted in parallel in the Clinical Investigation Center Plurithematic (CIC-P)1433 of Nancy (the study coordinating center) by the general practitioners investigators of the CIC-P.

The main purpose of the study is to determine the factors associated with the rate of patients remaining normotensive one year after stopping their antihypertensive monotherapy or low dose dual therapy:

* white coat hypertension
* primary diagnosis by home blood pressure measurements (HBPM) /ambulatory blood pressure measurements (ABPM) /clinical measure
* initial blood pressure level
* compliance
* therapeutic class versus others
* age
* gender
* weight variation
* modification of lifestyle
* concomitant treatments and associated substances
* ...

The primary endpoint will be the rate of normotensive patients at one year (i.e. HBPM values <135/85 mmHg).

DETAILED DESCRIPTION:
HBPM should be performed by the patients twice a day for 7 consecutive days before each visit (ESH protocol), using a device clinically tested (ESH/international protocol).

At baseline (visit 1), for the patients included, the antihypertensive treatment will be stopped in 3 consecutive days (half dose then interruption), over a maximum period of 12 months corresponding to the length of the participation and the monitoring of the patients.

Follow-up visits at day 30 (visit 2), day 90 (visit 3), day 180 (visit 4), day 270 (visit 5) and day 360 (visit 6). Will be performed at each visit:

* Calculation of the average of HBPM values by the investigator
* Measurements of office blood pressure (average of 3 consecutive measurements)
* SF 36 scale at baseline (visit 1) and day 360 (visit 6)
* During follow-up, the investigator will be free at any time to reintroduce an antihypertensive treatment if the average of HBPM values is greater than or equal to 135/85 mmHg on two consecutive visits, or greater than or equal to 155/95 mmHg regardless of the visit and regardless of the office blood pressure level.

At the end of study, the recovery of an antihypertensive treatment by the patients will be left to the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patient above 18 years old.
* Grade I hypertension at diagnosis.
* Hypertension diagnosed and treated (whatever is its seniority and for at least 6 months) by antihypertensive drug.
* Controlled hypertension (Clinical BP < 140/90 mmHg) or uncontrolled hypertension (Clinical BP > or equal to 140/90 mmHg) without modification of treatment for at least 6 months, by a monotherapy or a low dose dual therapy.
* HBPM values < 135/85mmHg (in order to exclude masked hypertension).
* Patient having signed the informed consent form.
* Patient affiliated to a national insurance scheme.

Exclusion Criteria:

* Personal cardiovascular history and/or necessity to take the antihypertensive treatment for another reason than hypertension (heart failure, migraine, peripheral arterial disease, coronary heart disease, stroke…).
* Target organ damage (evidence of ventricular hypertrophy by ECG or cardiac echography and/or proteinuria and/or pathological micro-albuminuria presence showing a nephropathy, in the last year).
* Poorly compliant patient, whose score of Girerd questionnaire is equal to or greater than 3.
* Existence of a progressive disease likely to impact on the life expectancy in a short term.
* Existence of a documented atrial fibrillation (contraindication of HBPM).
* Patient under a legal protection measure.
* Chronic alcohol or drug abuse, regular intake of vasopressor effect substances (licorice,cocaine,...).
* Current known pregnancy or project of pregnancy within one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2015-03-10; Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
The rate of normotensive patients at 1 year (i.e HBPM <135/85 mmHg) | At 12 months after antihypertensive treatment interruption

SECONDARY OUTCOMES:
The rate of normotensive patients at 3 months (i.e HBPM <135/85 mmHg) | At 3 months after antihypertensive treatment interruption
The rate of normotensive patients at 6 months (i.e HBPM <135/85 mmHg) | At 6 months after antihypertensive treatment interruption
The rate of normotensive patients at 9 months (i.e HBPM <135/85 mmHg) | At 9 months after antihypertensive treatment interruption
Evolution of the quality of life scale (part of SF36) | Change from baseline to 12 months after antihypertensive treatment interruption

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc BOIVIN, MD, PhD, Principal Investigator — Centre d'Investigation Clinique Plurithématique/INSERM/CHU de Nancy
Locations (24):
- France (24):
  - Cabinet de groupe Dr Birgé, Boulay
  - Cabinet de groupe Dr BAUDOIN, Bouzonville
  - Cabinet de groupe Dr Gries, Dettwiller
  - Cabinet du Dr Di Patrizio, Dombasle-sur-Meurthe
  - Cabinet médical Dr Bouché, Dombasle-sur-Meurthe
  - Cabinet médical du Dr Chevillard, Dombasle-sur-Meurthe
  - Maison de santé Dr Millet-Malingrey, Gondrecourt-le-Château
  - Maison de Santé Pluridisciplinaire de GROSTENQUIN, Grostenquin
  - Cabinet de groupe Dr Rougerie, Hatten
  - Cabinet du Dr Plane, Jarville-la-Malgrange
  - Cabinet médical prof Boivin, Laxou
  - Cabinet du Dr LARQUE, Le Palais-sur-Vienne
  - Cabinet de groupe Dr Faure Christian, Limoges
  - Cabinet Dr Bleynie, Limoges
  - Cabinet du Dr Poyeton, Neufchâteau
  - Cabinet Dr Delage, Nexon
  - Cabinet de groupe en pôle de santé, Revigny-sur-Ornain
  - Cabinet de groupe Dr Masson,, Rémilly
  - Cabinet du Dr Louyot-Keller, Saint-Avold
  - Cabinet médical du Dr Carrier, Saint-Max
  - Maison de Santé du Neuhof, Strasbourg
  - cabinet de groupe Dr Steyer, Talange
  - Centre d'Investigation Clinique module plurithématique 1433 Inserm/CHRU de Nancy, Vandœuvre-lès-Nancy
  - cabinet du Dr Gerard, Vicherey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boivin JM, Ferreira JP, Lopez-Sublet M, Duarte K, Zannad F, Rossignol P, Girerd N. Stopping antihypertensive Treatment amOng hypertensive patients in Primary care: The STOP-Trial. Eur J Prev Cardiol. 2025 Aug 21:zwaf511. doi: 10.1093/eurjpc/zwaf511. Online ahead of print. PMID 40838798